CLINICAL TRIAL: NCT00799032
Title: Assessment of The Latest Non-Thrombogenic Angioplasty Stent (ATLANTA): Prospective, First in Man, Non-Randomized, Single Center for Patients With Documented Myocardial Ischemia Undergoing PCI
Brief Title: The ATLANTA First in Man Study of the Catania Stent
Acronym: ATLANTA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CeloNova BioSciences, Inc. (Industry)
Responsible Party: Corrado Tamburino, MD, PhD, Ferrarotto Hospital, University of Catania
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-PC-002
Record Dates: First submitted 2008-11-25; First posted 2008-11-27 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stent (Other): Catania Stent
  Interventions: Device: PCI

INTERVENTIONS:
Device: PCI — coronary stent implantation
  Other Names: Catania Stent

SUMMARY:
To evaluate the short-term and mid-term safety and efficacy of the Catania coronary stent for the treatment of up to two de novo lesions in native coronary arteries.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, first-in-man single center study. The study requires a 55 patients with documented myocardial ischemia undergoing PCI.

ELIGIBILITY:
Inclusion Criteria:

* Lesion length ≤ 20 mm
* Vessel size ≥ 2.5 ≤ 3.5 mm

Exclusion Criteria:

* Life expectancy < 1 year
* Left ventricular ejection fraction (LVEF) <30%
* Anti-thrombotic drug intolerance

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Procedural success, Target Lesion Revascularization, Target Vessel Revascularization, Stent Thrombosis, Cardiac death, fatal/non fatal MI | In Hospital

SECONDARY OUTCOMES:
Any death, cardiac death, stent related fatal / non fatal Myocardial Infarction, Target Lesion Revascularization, Target Vessel Revascularization, Stent Thrombosis, Binary Restenosis | 1 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Corrado Tamburino, MD, Principal Investigator — Ferrarotto Hospital, University of Catania
Locations (1):
- Ferrarotto Hospital, Catania, Sicily, Italy